CLINICAL TRIAL: NCT01950546
Title: Nanosilver Fluoride: a Microbiological and Clinical Trial
Brief Title: Nanosilver Fluoride to Prevent Dental Biofilms Growth
Acronym: NSFCT
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: University of Pernambuco (Other)
Collaborators: Coordenação de Aperfeiçoamento de Pessoal de Nível Superior. (Other Government)
Responsible Party: Principal Investigator, Priscila Lima de Luna Freire, Msc, School of Dentistry, University of Pernambuco,, University of Pernambuco
Allocation: Not Applicable | Model: Single Group | Masking: Double | Purpose: Treatment
Other Study IDs: FOP01
Record Dates: First submitted 2013-09-16; First posted 2013-09-25 (Estimated); Last update posted 2015-06-10 (Estimated); Status verified 2015-06

CONDITIONS: Dental Caries
Keywords: silver nanoparticles; antimicrobial activity; toxicity; biofilm; cariostatic agents
MeSH Terms: conditions — Dental Caries | interventions — colloidal silver

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- Nanosilver fluoride (Experimental): This product is a solution composed of: 390 mg / ml 9nm silver nanoparticles ;21 mg / ml chitosan ; 22 mg / ml NaF.The cariostatic agent, nanosilver fluoride, was formulated in a similar way to silver diamine fluoride, so that this new formulation contained 5% nanosilver fluoride, while commercial diamine silver fluoride contains 30% silver fluoride. It will be applied once with a microbrush on tooth surfaces to check if it prevents the growth of S. mutans biofilms on dental surfaces.
  Interventions: Drug: nanosilver fluoride

INTERVENTIONS:
Drug: nanosilver fluoride — The product will be applied in the volunteers in the morning, before the first class, in relative isolation, made with cotton rolls and Vaseline to protect the soft tissue. It will apply 30mg of the product with microbrush, previously standardized in a pilot study on cervical vestibular surfaces of incisors and canines healthy, on a total of 8 teeth, 4 upper and 4 lower. After a period of 7 days,the cervical dental biofilms will be collect, third on the buccal surfaces of incisors and / or canines upper and lower, with the aid of sterile spatulas.
  Other Names: silver nanoparticles

SUMMARY:
This study aims to evaluate the effectiveness of nanosilver fluoride for controlling the growth of S. mutans present in dental plaque of children.

DETAILED DESCRIPTION:
The product will be apllied on cervical vestibular surfaces of incisors and canines healthy, with a total of 8 teeth, 4 upper and 4 below. Children will be instructed not to ingest any liquid or food within two hours after application. After a period of 7 days will be carried biofilm colect of cervical dental surfaces of incisors and / or canines upper and lower, with the aid of sterile spatulas. This material will be packaged in pre-weighed microfuge tubes containing 1.5 ml of buffered saline solution (0.9% sodium chloride), and transported under refrigeration immediately to the laboratory where analysis will be performed and the S. mutans colonies will be counted. The biofilm collect and posterior laboratorial analysis will be performed weekly.

ELIGIBILITY:
Inclusion Criteria:

* Have at least 4 upper teeth and 4 lower teeth deciduous;systemic health satisfactory; did not use antibiotics or nonsteroidal anti-inflammatory within one month before or during the study;do not use any other forms of chemical control of biofilm during the study period;not being a user of orthodontic devices or dentures;

Exclusion Criteria:

* Presenting oral lesions, supragingival calculus and severe malocclusion.

Ages: 5 Years to 6 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Enrollment: 30 (Actual)
Dates: Start 2014-09; Primary Completion 2014-12 (Actual); Study Completion 2015-01 (Actual)

PRIMARY OUTCOMES:
Initial biofilm collecting before applying the product and after nanosilver fluoride application. | one week
  The initial dental biofilm collection will be conducted to count colony-forming units of S. mutans and then the product will be applied on these dental surfaces after the collect. After one week, a new collect will be performed and the colony-forming units of S. mutans will be counting to compare with the initial.

SECONDARY OUTCOMES:
Evaluation of effectiveness of nanosilver fluoride on bacterial growth in the dental biofilm | two weeks
  Collection of dental biofilm will be performed after two weeks of product application and colony count will be performed in the laboratory.

OTHER OUTCOMES:
Collection of dental biofilm will after four weeks of product application. | Four weeks
  Collection of dental biofilm will be performed after four weeks of product application and colony count will be performed in the laboratory.
Collection of dental biofilm after eight weeks of product application | Eight weeks
  Collection of dental biofilm will be performed after eight weeks of product application and will be compared with the initial score of S. mutans colony forming units.

CONTACTS AND LOCATIONS:
Overall Officials: Aronita Rosenblatt, PhD, Study Director — UPE
Locations (1):
- Escola Municipal Anita Trigueiro do Valle, João Pessoa, Paraíba, Brazil